CLINICAL TRIAL: NCT04585048
Title: The Efficacy of Integrated Behavioral Therapy for Selective Mutism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, alan apter, Prof. Alan Apter, Rabin Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0210-15-RMC
Record Dates: First submitted 2019-02-10; First posted 2020-10-14 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Selective Mutism
MeSH Terms: conditions — Mutism

STUDY DESIGN:
Intervention Model Description: waiting list vs. treatment phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- waiting list (No Intervention): waiting list
- treatment (Experimental): treatment with the Integrated Behavioral Therapy fo Selective Mutism
  Interventions: Behavioral: Integrated Behavioral Therapy for Selective Mutism

INTERVENTIONS:
Behavioral: Integrated Behavioral Therapy for Selective Mutism — Cognitive Behavioral treatment including 24 weekly sessions
  Arms: treatment

SUMMARY:
This study examines the efficacy of the Integrated Behavioral Therapy for Selective Mutism protocol (Bergman et al., 2013). Participants are 60 children, aged 4-8 years, diagnosed with Selective Mutism (SM). The level of SM symptoms is assessed during first arrival to the SM unit of Schneider Children's Medical Center of Israel (Intake), at the first treatment session, at sessions 12, and at the end of treatment.

A secondary aim of this study is to assess the contribution of parent's characteristics (anxiety and depression levels, parenting style) to the childrens' SM symptoms level and to treatment achievements.

DETAILED DESCRIPTION:
All study procedures have been approved by the Institutional Review Board of Schneider Children's Medical Center of Israel. Participants are recruited from the Selective Mutism unit at Schneider Children's Medical Center of Israel, during their first visit to the clinic. Both parents of eligible children sign informed consents. Each child is evaluated by a clinical psychologist, using a semi-structured interview (ADIS), designed to diagnose the child and to determine the level of symptom severity. The parents who are identified as the main-caregiving, complete questionnaires assessing the child's levels of SM symptoms and social anxiety (SMQ, SASC), the parents' levels of social anxiety (LSAS, SPIN) and depression (BDI), parent's authority style (PAQ), parental accommodation (FASA) and parental playfulness (PPQ). The child's teacher completes questionnaires assessing the child's SM levels (SSQ). Participants are than assigned either to the treatment or the waiting list group (by chance). The assessment of SM levels is repeated in both groups at 1 week from baseline, 12 weeks from baseline, and 24 weeks from baseline. participants of the waiting list group will commence treatment following the 24 weeks waiting period.

ELIGIBILITY:
Inclusion Criteria:

* Selective Mutism diagnosis (DSM-5)
* age 4-8 years

Exclusion Criteria:

* Autism Spectum Disorder
* Psychotic disorder
* Commenced other psychiatric or psychological treatment at the last month

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-05-14 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Selective Mutism Questionnaire | baseline, 1 week from baseline, 12 weeks from baseline, 24 weeks from baseline
  The change in parent's and teacher's report on child's selective Mutism symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Maayan shorer, PhD, Study Director — Schneider Children's Medical Center, Israel
Locations (1):
- Schneider Childrens' Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No